CLINICAL TRIAL: NCT05721417
Title: Long-term Outcomes of Isolated Tricuspid Valve Surgery According to Preoperative Clinical and Functional Staging
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: LOITAPF
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tricuspid valve surgery — Surgical treatment of tricuspid regurgitation, that may be performed by repair or replacement

SUMMARY:
Tricuspid regurgitation (TR) was identified as an independent prognostic factor associated with excess mortality and morbidity, independent of left ventricular (LV) function and pulmonary hypertension. Isolated tricuspid surgery has been performed for a long time in a few selected cases, however in recent years several studies have underlined how the poor outcomes described for isolated tricuspid valve surgery seem to be related to the baseline characteristics of the patients and to late referral for surgical treatment rather than the intervention itself. To facilitate patient screening, a new clinical and functional TR staging system has recently been proposed. This classification, which evaluates the progression of morphological variations of the tricuspid valve and right ventricle (RV) in association with the onset of symptoms, identifies several parameters and factors that can be useful for a better stratification of surgical risk. Rather than simply assessing the degree of TR, this new staging mechanism also focuses on symptoms, RV remodeling and function, medical therapy, and right heart failure hospitalizations.

Investigators previously focused on the short-term (mainly hospital) outcomes of patients undergoing isolated surgery for severe TR, who were classified at baseline according to this clinical and functional staging system. Results showed that a more comprehensive classification reflects the population and hospital outcomes of surgically treated patients with isolated TR.

The purpose of this study is to ultimately evaluate long-term outcomes of this patients population and estimate the impact of baseline staging on long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Affected by severe tricuspid regurgitation (TR), both of degenerative and functional etiology and;
* Patients underwent isolated surgery, either repair or replacement, of the tricuspid valve
* Patients operated on at theCardiac Surgery Department of San Raffaele Hospital from May 2004 to May 2020.

Exclusion Criteria:

- Patients with non-isolated tricuspid valve surgery (concomitant surgery on other valves).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by severe TR, degenerative or functional, requiring isolated (not concomitant with other valvular procedures) repair or replacement of the tricuspid valve
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 17 years
Reoperation for TR recurrency | Up to 17 years
Right heart failure hospitalization incidence | Up to 17 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No